CLINICAL TRIAL: NCT01726985
Title: Model for Heart Failure ExAcerbation Reduction Trial - "Model HEART"
Brief Title: Model for Heart Failure ExAcerbation Reduction Trial
Acronym: HEART
Status: Completed | Type: Observational
Sponsor: Cleveland Clinic Florida (Other)
Responsible Party: Sponsor
Organization: The Cleveland Clinic (Other)
Other Study IDs: 121368
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2012-11

CONDITIONS: Acute on Chronic Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients hospitalized with CHF: Patients hospitalized with CHF Parameter Based Clinical Disposition
  Interventions: Other: Parameter Based Clinical Disposition

INTERVENTIONS:
Other: Parameter Based Clinical Disposition — Parameter Based Clinical Disposition'
  Physicians will initiate / titrate medications and obtain consults as usual but are highly encourage to keep patients in the hospital until at least 2 of the following 3 criteria are met:
  * NT-ProBNP reduction of > 23% from peak value during admission
  * Fluid Reduction of > 1.3L (orders for I/O q8h required)
  * Serum Sodium of > 135 mmol/L the day of planned discharge

SUMMARY:
Heart failure is the leading cause of hospitalizations and readmissions in the United States and is a tremendous economic strain on our healthcare system. There is currently, based on national averages, a 30% readmission rate and 10% mortality rate within 3 months of being hospitalized for heart failure. Retrospective studies have shown benefit to using biomarkers such as BNP to guide inpatient heart failure management. Our own CCF retrospective study showed that decreasing NT-ProBNP by 23%, making patients fluid negative by more than 1.3L, and discharging patients with serum sodium above 135 reduces readmission rates significantly. The purpose of this study is to prospectively use the above mentioned goals in the treatment of heart failure in order to reduce heart failure readmission and mortality rates.

DETAILED DESCRIPTION:
All HF patients admitted to CCF will receive a short consent form. The study will enroll patients for one year. Physicians will initiate / titrate medications and obtain consults as usual but are highly encourage to keep patients in the hospital until at least 2 of the 3 (above mentioned) criteria are met. Physicians will receive a copy of consent forms, educational bulletins, and discharge forms (as described in the Physician Education document which is attached to this application). Log-rank test will be used to compare groups. Chi-Square will be used to compare prospective patients with retrospective controls (obtained in 2010).

ELIGIBILITY:
Inclusion Criteria:

* Must have either Acute on Chronic Heart Failure or Chronic Heart Failure regardless of presenting/primary complaint

To fulfill CHF Dx, MUST have 2+ of the following:

* Clinical: Dyspnea, orthopnea, PND, edema, S3, rales, improve w diuretics
* Radiographic: Pulm venous congestion, pleural effs, cardiomegaly
* Lab: NT pro BNP > 1000

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18 and over hospitalized at Cleveland Clinic Florida with diagnosis of CHF.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2012-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Hospital Readmission for CHF | up to 1 year

SECONDARY OUTCOMES:
CHF Mortality | 90 days, 180 days, 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: Marlow Hernandez, Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No